CLINICAL TRIAL: NCT01366573
Title: A Randomised, Double-Blind, Single-Dose, Four-Period Cross-Over Study to Determine the Effects of Alcohol on the Pharmacokinetics and Pharmacodynamics of GSK1521498 in Healthy Subjects
Brief Title: GSK1521498 Alcohol Interaction Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: University of Cambridge (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 115256
Record Dates: First submitted 2011-05-12; First posted 2011-06-06 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Alcoholism
Keywords: Pharmacokinetics; mu-opioid receptors; Addiction; Pharmacodynamics; Alcohol
MeSH Terms: conditions — Alcoholism; Behavior, Addictive | interventions — N-((3,5-difluoro-3'-(1H-1,2,4-triazol-3-yl)-4-biphenylyl)methyl)-2,3-dihydro-1H-inden-2-amine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- GSK1521498 & alcohol (Experimental): GSK1521498 20 mg and alcohol (0.5g/kg ethanol mixed with orange juice)
  Interventions: Drug: GSK1521498
- GSK1521498 & orange juice (Experimental): GSK1521498 20 mg and orange juice approximately matching alcoholic beverage for volume and colour
  Interventions: Drug: GSK1521498
- Placebo & alcohol (Experimental): Placebo and alcohol (0.5g/kg ethanol mixed with orange juice)
  Interventions: Other: Placebo
- Placebo & orange juice (Placebo Comparator): Placebo and orange juice approximately matching alcoholic beverage for volume and colour
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: GSK1521498 — GSK1521498 20 mg administered with alcohol to determine PK/PD interactions
  Arms: GSK1521498 & orange juice; GSK1521498 & alcohol
Other: Placebo — Placebo
  Arms: Placebo & alcohol; Placebo & orange juice

SUMMARY:
The aim of the study is to assess the safety and tolerability of GSK1521498 in combination with alcohol and to determine the amount of GSK1521498 and alcohol in your blood after you have been given these together. The study will also determine whether GSK1521498 will have an effect on alcohol liking and consumption.

DETAILED DESCRIPTION:
The study is to test a new drug which may be used for treating alcohol addiction. The drug works by inhibiting the effects of messenger molecules called opioids. These opioids are naturally produced within the human body, and are involved in controlling how much alcohol we drink and the pleasure we get from drinking alcohol. We believe that GSK1521498 might be effective in the treatment of alcohol addiction because it is well known that drugs working on similar binding sites in the brain reduce the pleasure we get from drinking alcohol. As alcohol can effect the way that a drug is metabolised in the body, The investigators need to determine that it is safe to take GSK1521498 in combination with alcohol. and to determine the amount of GSK1521498 and alcohol in your blood after you have been given these together. The study will also determine whether GSK1521498 will have an effect on alcohol liking and consumption.

ELIGIBILITY:
Inclusion Criteria:

* healthy male or female between 21 and 55 years of age inclusive.
* within 20% normal weight for height and body build.
* A female subject of child-bearing potential must use one of the contraception methods listed in the protocol prior to the start of the study until at least 14 days after receiving the last dose of study medication.
* Male subjects must agree to use one of the contraception methods listed in the protocol from the time of the first dose of study medication until at least 5 days after receiving the last dose of study medication.
* History of regular alcohol consumption within 6 months of study.
* No recent changes in patterns of alcohol consumption.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

* A positive test for HIV, Hep B or Hep C.
* Current or chronic history of liver disease.
* Current or chronic history of neurological disorders.
* Subjects with previous or current psychiatric history.
* Past history of DSM-IV alcohol dependence or abuse.
* Binge drinking more than once a week (>5 standard drinks in one session is a binge).
* Currently trying to quit alcohol.
* Positive urine screen for amphetamines, barbiturates, cocaine, opiates, cannabinoids or bezodiazepines at screening.
* Regular consumption of >450mg caffeine per day (an average cup contains about 75mg).
* Heavy smokers, defined as those who smoke >10 cigarettes a day. Also those who cannot abstain during the admission period.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 14 days prior to the first dose of study medication.
* Pregnant or lactating females.
* QTcB or QTcF >450msec.
* Participated in a clinical trial and has received an investigational product within 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product.
* Where participation in the study would result in donation of blood or blood products in excess of 500mL within a 56 day period.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2011-05-13 (Actual); Primary Completion 2011-09-16 (Actual); Study Completion 2011-09-16 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic interaction | GSK1521498 PK sampling; pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 9, 12, 13, 24, 48 and 72 hr post-dose.
  AUC and Cmax of GSK1521498 and alcohol

SECONDARY OUTCOMES:
Safety: adverse events, vital signs, ECGs, physician/nurse observations, safety lab tests, mood assessments | 3 Months
Neurological assessments including Purdue Pegboard test | 3 Months

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Results for study 115256 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/115256?search=study&study_ids=115256#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 115256 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 115256 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 115256 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 115256 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 115256 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 115256 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 115256 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register